CLINICAL TRIAL: NCT04379440
Title: Geriatric Population COVID-19 Syndromic Characteristics and Clinical Outcomes: a Multi-setting, Multi-domain Observational Study (GEROCOVID Observational)
Brief Title: Geriatric Population COVID-19 Observational Study (GEROCOVIDobs)
Acronym: GEROCOVIDobs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Raffaele Antonelli Incalzi (Other)
Collaborators: Italian Society of Gerontology and Geriatrics (Unknown); BLUECOMPANION FRANCE (Unknown); BLUECOMPANION LTD (Unknown)
Responsible Party: Sponsor-Investigator, Raffaele Antonelli Incalzi, Full Professor in Internal Medicine, Director of Geriatrics Department and Acting Director of Chronic Diseases Department, Campus Bio-Medico University
Organization: Campus Bio-Medico University (Other)
Other Study IDs: GC01-Obs
Record Dates: First submitted 2020-05-03; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: Coronavirus Electronic Registry Geriatrics Best Practices
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- " Acute Ward Patients " care setting cohort: Acute Ward Hospitalised patients with suspected or known SARS-CoV-2 infection
- " Nursing Homes (RSA) " care setting cohort: Nursing Home Resident Older Adult suffering from Suspected or known SARS-CoV-2 infection
- " Home and Outpatients' Care " cohort: Outpatients at risk of SARS-CoV-2 infection
- " Dementia Outpatients " cohort: Outpatients suffering from Dementia according to NIA-AA criteria, at risk of SARS-CoV-2 infection and on Treatment with anti-cholinesterase- dugs and/or anti-psychotics
- " At home " cohort: Outpatients at risk of SARS-CoV-2 infection
- " Outcomes " cohort: Age≥65 years as target population Hospitalised patients diagnosed with SARS-CoV-2 infection

SUMMARY:
The GeroCovid e-Registry is a European de-identified clinical data electronic registry of geriatric patients at risk or suffering from COVID-19 (suspected and confirmed cases) observed since 1st March 2020 in the participating investigational sites.

DETAILED DESCRIPTION:
Older adults (≥ 65 years) and pre-geriatric population (≥60 years and <65 years) are the ones most at risk from complications of COVID-19, including increased mortality, possibly in relationship with their comorbidity and frailty status.

The GeroCovid e-registry is intended to track Covid-19 pandemic impact on the general geriatric population and on age/care-setting related sub-populations.

The analysis of results is expected to facilitate the adoption of optimal standard of geriatric care during the pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Applying only to the " Acute Ward Patients " cohort:

   1. Hospitalised patients
   2. Suspected or known SARS-CoV-2 infection
2. Applying only to the "Nursing Homes (RSA)" cohort:

   1. Nursing Home Resident Older Adults
   2. Suspected or known SARS-CoV-2 infection
3. Applying only to the" Home and outpatients' care " cohort:

   a. Outpatients at risk of SARS-CoV-2 infection
4. Applying only to the" Dementia outpatients " cohort:

   1. Outpatients suffering from dementia according to NIA-AA criteria
   2. At risk of SARS-CoV-2 infection
   3. Ongoing treatment with anti-cholinesterase- dugs and/or anti-psychotics
5. Applying only to the" At home " cohort:

   a. Outpatients at risk of SARS-CoV-2 infection
6. Applying only to the " Outcomes " cohort:

   1. Age≥65 years
   2. Hospitalised patients diagnosed with SARS-CoV-2 infection

Exclusion Criteria:

1. Lack of a signed Informed Consent if the patient received and understood the information about the study.
2. Lack of a signed declaration by the responsible physician stating that no explicit opt-out advanced directives by the subject were known to be in place at the moment of inclusion if it had been impossible to inform the patient due to her/his state of consciousness and/or awareness of disease condition.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sequentially observed cases since the start of the registry at the Investigational Centre. The registry can be started on 1st March 2020 at the earliest.
  Older adults theoretically at risk of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Health status (WHO classification) | 60 days or less in case of early termination
  Change of health status according to WHO classification versus baseline after 60 days, or after any interval (last performed observation) in the event of early study termination (whole sample).
Incidence of Serious Adverse Events | 60 days or less in case of early termination
  Incidence and duration of hospitalisation, incidence of Death and other Serious Adverse Events;

SECONDARY OUTCOMES:
COVID-19 prevalent symptoms at onset | Day0
  Most frequent symptoms coded according MedDRA dictionary as reported at hospital admission
COVID-19 Prognostic Factors | Day0
  Most frequent chronic diseases (coded according MedDRA dictionary) as reported at hospital admission per Outcome (death; Serious Adverse Event other than death).
Incidence of COVID-19 in the RSA cohort | 60 days or less in case of early termination
  Incidence of COVID-19 in the Nursing Homes (RSA) cohort per specific preventive measures application
Affective/mood state change from baseline in the " At home " cohort | 60 days or less in case of early termination
  Affective/mood state measured by the Geriatric Depression Scale 5-items (GDS-5) change from baseline; the GDS-5 ranges from 0 to 5, with scores>2 suggesting depression
Cognitive function in the "Dementia" and "At home " cohorts | 60 days or less in case of early termination
  Mini Mental State Exam ( MMSE) change from baseline; the MMSE range from 0 to 30, with scores of 26 or higher being traditionally considered normal. Scores less than 9 generally indicate severe impairment, while scores between 10 and 20 indicate moderate dementia.
Daily Life Function in the "Dementia" and "At home " cohorts | 60 days or less in case of early termination
  Activities of Daily Life rating scale ( ADL) change from baseline; the ADL range from 6 to 0, 6 = High (patient independent) 0 = Low (patient very dependent)
Instrumental Daily Life function in the "Dementia" and "At home " cohorts | 60 days or less in case of early termination
  Instrumental Activities of Daily Life rating scale ( iADL) change from baseline; the iADL summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women and 0 through 5 for men to avoid potential gender bias.
Residual signs and symptoms in the " Outcomes " cohort | 60 days or less in case of early termination
  Prevalence and pattern of residual signs and symptoms in the " Outcomes " cohort
Incidence of outcomes in the " Outcomes " cohort per Frailty Status | 60 days or less in case of early termination
  Incidence of Death, Hospitalisation, Hospitalisation days, number of Serious Adverse Events) per Frailty Status at baseline (Fried's anamnestic criteria, adapted)
Incidence of outcomes in the " Outcomes " cohort per Comorbidity burden at baseline | 60 days or less in case of early termination
  Incidence of outcomes (Death, Hospitalisation, Hospitalisation days, number of Serious Adverse Events) per Comorbidity Burden at baseline (CIRS)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Antonelli Incalzi, M.D., Principal Investigator — Policlinico Campus Bio-Medico
Locations (7):
- Italy (7):
  - RSA La Quiete, Castiglione Cosentino, Calabria
  - ASP Catanzaro, Catanzaro Lido, Calabria
  - AOU Ferrara, Ferrara, Emilia-Romagna
  - Policlinico Campus Bio-Medico, Rome, Roma
  - AOU Careggi, Florence, Tuscany
  - AOU Pisana Geriatria, Pisa, Tuscany
  - Ospedale di Comunita' ULSS 6 Euganea- COVID Center, Camposampiero, Veneto

REFERENCES:
- [Derived] Gareri P, Trevisan C, Abbatecola AM, Malara A, Incalzi RA. Efficacy of OM-85 in Recurrent Respiratory Tract Infections. Rev Recent Clin Trials. 2023;18(3):223-227. doi: 10.2174/1574887118666230518112806. PMID 37202893
- [Derived] Trevisan C, Remelli F, Fumagalli S, Mossello E, Okoye C, Bellelli G, Coin A, Malara A, Gareri P, Monzani F, Del Signore S, Zia G, Antonelli Incalzi R, Volpato S; GeroCovid Acute Ward Working Group. COVID-19 as a Paradigmatic Model of the Heterogeneous Disease Presentation in Older People: Data from the GeroCovid Observational Study. Rejuvenation Res. 2022 Jun;25(3):129-140. doi: 10.1089/rej.2021.0063. Epub 2022 Jun 6. PMID 35570723
- [Derived] Okoye C, Finamore P, Bellelli G, Coin A, Del Signore S, Fumagalli S, Gareri P, Malara A, Mossello E, Trevisan C, Volpato S, Zia G, Monzani F, Incalzi RA. Computed tomography findings and prognosis in older COVID-19 patients. BMC Geriatr. 2022 Mar 1;22(1):166. doi: 10.1186/s12877-022-02837-7. PMID 35227201
- [Derived] Fumagalli S, Trevisan C, Del Signore S, Pelagalli G, Fumagalli C, Herbst A, Volpato S, Gareri P, Mossello E, Malara A, Monzani F, Okoye C, Coin A, Bellelli G, Zia G, Ungar A, Ranhoff AH, Antonelli Incalzi R; GeroCovid Working Group. Atrial fibrillation and COVID-19 in older patients: how disability contributes to shape the risk profile. An analysis of the GeroCovid registry. Aging Clin Exp Res. 2022 Jan;34(1):249-256. doi: 10.1007/s40520-021-02008-5. Epub 2021 Oct 30. PMID 34716570
- [Derived] Trevisan C, Del Signore S, Fumagalli S, Gareri P, Malara A, Mossello E, Volpato S, Monzani F, Coin A, Bellelli G, Zia G, Ranhoff AH, Antonelli Incalzi R; GeroCovid Working Group. Assessing the impact of COVID-19 on the health of geriatric patients: The European GeroCovid Observational Study. Eur J Intern Med. 2021 May;87:29-35. doi: 10.1016/j.ejim.2021.01.017. Epub 2021 Jan 31. PMID 33573885